CLINICAL TRIAL: NCT02676401
Title: An Extended Treatment Study of MT-3995 in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT-3995-J06
Record Dates: First submitted 2016-02-01; First posted 2016-02-08 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MT-3995 Low (Experimental)
  Interventions: Drug: MT-3995 Low
- MT-3995 Middle (Experimental)
  Interventions: Drug: MT-3995 Middle
- MT-3995 High (Experimental)
  Interventions: Drug: MT-3995 High

INTERVENTIONS:
Drug: MT-3995 Low
  Arms: MT-3995 Low
Drug: MT-3995 Middle
  Arms: MT-3995 Middle
Drug: MT-3995 High
  Arms: MT-3995 High

SUMMARY:
This study aims to evaluate the safety and efficacy of MT-3995 administered over the longer term, following MT-3995-J05 study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for participation before the completion of MT-3995-J05 Study
* Completion of MT-3995-J05 study

Exclusion Criteria:

* UACR of ≥300 mg/g Cr with an increase of ≥30% in MT-3995-J05 Study
* Symptomatic and clinically significant hypotension
* QT prolongation or torsades de pointes
* New York Heart Association (NYHA) Class III or IV heart failure
* Patients who are judged to be unsuitable for participation based on their safety profile in MT-3995-J05 Study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2016-02; Primary Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Adverse events | From baseline to 28 weeks

SECONDARY OUTCOMES:
Change from baseline in Urine Albumin to Creatinine Ratio (UACR) | baseline and Week 28

CONTACTS AND LOCATIONS:
Locations (1):
- Touei Hospital, Hokkaido, Japan

REFERENCES:
- [Derived] Wada T, Inagaki M, Yoshinari T, Terata R, Totsuka N, Gotou M, Hashimoto G. Apararenone in patients with diabetic nephropathy: results of a randomized, double-blind, placebo-controlled phase 2 dose-response study and open-label extension study. Clin Exp Nephrol. 2021 Feb;25(2):120-130. doi: 10.1007/s10157-020-01963-z. Epub 2020 Sep 24. PMID 32974732